CLINICAL TRIAL: NCT06929169
Title: Cardiovascular Effects of SGLT2 Inhibitors in Hemodialysis Patients: A Phase 2 Randomized Study
Acronym: SGLT2-HD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maximo Agustin Schiavone (Other)
Responsible Party: Sponsor-Investigator, Maximo Agustin Schiavone, Principal Investigator and Sponsor-Investigator, CEMIC, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Organization: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIISA BA: 8767
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: SGLT2 Inhibitors; Hemodialysis; Cardiac MRI; Ventricular Remodeling; Heart Failure with Preserved Ejection Fraction; Myocardial Fibrosis; Cardiovascular Disease; Chronic Kidney Disease
MeSH Terms: conditions — Ventricular Remodeling; Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this arm will continue receiving standard hemodialysis treatment, including all routine medical care, medications, and monitoring as per institutional protocols. They will not receive an SGLT2 inhibitor.
- Drug: iSGLT2 (Experimental): Participants in this arm will receive a sodium-glucose cotransporter 2 inhibitor (SGLT2i) once daily by oral administration, in addition to standard hemodialysis care. The specific agent (e.g., dapagliflozin or empagliflozin) and dose will be selected based on safety data and existing recommendations for patients with end-stage renal disease on dialysis. The intervention will be administered for 12 months. Participants will undergo cardiovascular monitoring, including cardiac MRI, echocardiography, and biomarker assessment at baseline, and months 3, 6, and 12. This arm is designed to evaluate the effects of SGLT2 inhibition on cardiac function, myocardial fibrosis, and intradialytic hypotension.
  Interventions: Drug: iSGLT2

INTERVENTIONS:
Drug: iSGLT2 — Participants randomized to the experimental arm will receive a once-daily dose of a sodium-glucose cotransporter 2 inhibitor (SGLT2i), administered orally, in addition to their standard hemodialysis care. The specific agent (e.g., dapagliflozin or empagliflozin) and dose will be selected based on safety data and clinical guidelines applicable to patients with end-stage renal disease (ESRD) on dialysis. The intervention will be maintained for 12 months. Dosing will be monitored by the research team to ensure tolerability and adherence. All patients in the experimental group will undergo comprehensive cardiovascular assessment, including serial cardiac MRI, echocardiography, and measurement of fibrosis-related biomarkers.
  This intervention differs from standard care by introducing a pharmacologic agent not routinely administered in the dialysis population, targeting cardiac remodeling, fibrosis, and intradialytic complications.
  Other Names: SGLT2 inhibitor
  Arms: Drug: iSGLT2

SUMMARY:
Patients with end-stage kidney disease (ESKD) on hemodialysis face an unacceptably high rate of cardiovascular complications, including heart failure, arrhythmias, and sudden cardiac death. Many of these outcomes are driven by diastolic dysfunction and cardiac fibrosis-conditions that are not adequately addressed by current therapies. SGLT2 inhibitors, originally developed for the treatment of type 2 diabetes, have demonstrated cardiovascular and renal protective effects across multiple patient populations, independent of glycemic control.

This Phase 2, randomized, controlled clinical trial will evaluate the safety and efficacy of SGLT2 inhibitors in patients undergoing maintenance hemodialysis. A total of 80 participants will be randomized to receive either an SGLT2 inhibitor or standard care for 12 months. The primary objective is to determine whether SGLT2 inhibitors improve cardiac function, reduce myocardial fibrosis, and decrease the incidence of intradialytic hypotension. Secondary endpoints include cardiovascular events, hospitalization, and all-cause mortality. The study will also assess changes in key biomarkers and perform advanced cardiac imaging to evaluate structural and functional outcomes.

This trial represents a novel and timely investigation into a class of medications with promising pleiotropic effects, potentially offering new therapeutic options for a high-risk, underserved population.

DETAILED DESCRIPTION:
This is a Phase 2, prospective, randomized, open-label, controlled study designed to assess the safety and efficacy of sodium-glucose cotransporter 2 inhibitors (SGLT2i) in patients with end-stage renal disease (ESRD) undergoing maintenance hemodialysis. Despite advances in renal replacement therapy, cardiovascular mortality remains the leading cause of death in this population, often due to heart failure with preserved ejection fraction (HFpEF), arrhythmic events, and myocardial fibrosis. Preclinical models and clinical data in non-dialysis populations suggest that SGLT2 inhibitors exert antifibrotic, anti-inflammatory, and mitochondrial-stabilizing effects that may ameliorate these pathophysiological processes.

A total of 80 eligible patients, aged 18-70 years and receiving online hemodiafiltration for at least 3 months, will be enrolled at Fresenius Medical Center - CEMIC Saavedra (Buenos Aires, Argentina). Participants will be randomized into two parallel groups (intervention vs. control) stratified by age, sex, and dialysis vintage. The intervention group will receive a once-daily SGLT2 inhibitor, while the control group will continue standard care.

Primary outcomes include the incidence and severity of intradialytic hypotension (defined by KDOQI 2020 and HEMO criteria), longitudinal changes in left ventricular mass index (LVMI), ejection fraction, myocardial fibrosis as assessed by cardiac MRI (T1/T2 mapping), and circulating pro-fibrotic biomarkers (e.g., FGF23, procollagen types I and III). Secondary endpoints include major adverse cardiovascular events (MACE), cardiovascular mortality, all-cause mortality, and cause-specific hospitalizations.

Comprehensive phenotyping will be conducted at baseline, months 3, 6, and 12. Assessments include echocardiography, cardiac MRI, 24-hour Holter monitoring, impedance cardiography, pulse wave velocity measurement, and detailed laboratory profiling. Data will be analyzed using appropriate parametric and non-parametric statistical tests, with multivariate regression and survival analysis techniques applied where relevant.

The study complies with ICH-GCP guidelines and the Declaration of Helsinki. The CEMIC institutional review board has granted ethical approval. Informed consent will be obtained from all participants prior to enrollment. The study is funded by institutional and investigator resources, with biomarker assays supported by the lead investigator through his research affiliations with CEMIC and Charité -Universitätsmedizin Berlin.

This study aims to address a critical unmet need in cardio-renal medicine and may lay the groundwork for future therapeutic strategies in dialysis-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years
* Diagnosed with end-stage renal disease
* Undergoing online hemodiafiltration for at least 3 months
* Able to provide written informed consent

Exclusion Criteria:

* Current immunosuppressive therapy
* Contraindication to cardiac MRI
* Known hypersensitivity or intolerance to SGLT2 inhibitors
* Participation in another interventional clinical trial
* History of diabetic ketoacidosis
* Active substance abuse
* Diagnosis of type 1 diabetes mellitus
* History of kidney transplantation
* Acute coronary event within 30 days before enrollment
* Current or recent treatment with an SGLT2 inhibitor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Mass Index (LVMI) | Baseline, Month 3, Month 6, and Month 12
  LVMI will be measured using cardiac MRI and/or echocardiography at baseline, and at months 3, 6, and 12. The primary outcome will be the change (Δ) in LVMI compared to baseline. Reductions in LVMI will be interpreted as a marker of reverse remodeling and reduced fibrosis.
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, Month 3, Month 6, Month 12
  LVEF will be measured by echocardiography at baseline and at months 3, 6, and 12. The primary outcome will be the change from baseline. Improvements will indicate enhancement in global systolic function.
Change in Myocardial Fibrosis as Assessed by Cardiac MRI | Baseline, Month 3, Month 6, Month 12
  Cardiac MRI with T1/T2 mapping will be performed at baseline, and at months 3, 6, and 12. Quantitative measures of myocardial fibrosis will be compared to baseline to assess changes over time.
Change in Pro-fibrotic Biomarkers (FGF23, Procollagen I and III) | Baseline, Month 3, Month 6, Month 12
  Blood levels of FGF23, procollagen type I, and procollagen type III will be measured at baseline and months 3, 6, and 12. The outcome is defined as the change from baseline. These biomarkers reflect myocardial fibrosis activity.
Incidence of Intradialytic Hypotension | Baseline through Month 12
  Includes new or worsening heart failure, confirmed myocardial infarction, stroke, or clinically significant arrhythmia. Events will be adjudicated based on clinical criteria.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | Baseline through Month 12
  Includes new or worsening heart failure, confirmed myocardial infarction, stroke, or clinically significant arrhythmia. Events will be adjudicated based on clinical criteria.
Cardiovascular Mortality | Baseline through Month 12
  Deaths due to cardiovascular causes, including sudden cardiac death, will be recorded and classified according to investigator assessment and clinical documentation.
All-Cause Mortality | Baseline through Month 12
  All deaths occurring during the study period will be recorded regardless of cause. Attribution (cardiac, non-cardiac, unknown) will be documented when possible.
Cause-Specific Hospitalizations | Baseline through Month 12
  Hospitalizations will be recorded and categorized as cardiovascular, infectious, AV-fistula-related, or other. Events will be assessed from enrollment through study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Castellaro, MD, MSc, Study Director — Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Locations (1):
- Fresenius Medical Care - CEMIC Saavedra, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided